CLINICAL TRIAL: NCT01039675
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Combination of GSK573719 and GW642444 in Subjects With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113120
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: long-acting beta2-receptor agonist; Safety and tolerability; pharmacodynamics; pharmacokinetics; long-acting muscarinic receptor antagonist; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK573719/GW642444 (Experimental)
  Interventions: Drug: 500mcg/25mcg once daily
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo once daily

INTERVENTIONS:
Drug: 500mcg/25mcg once daily — GSK573719/GW642444
  Arms: GSK573719/GW642444
Drug: Placebo once daily — Inactive, excipients only
  Arms: Placebo

SUMMARY:
The study will evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of the combination of inhaled GSK573719 and GW64244 compared to placebo, in subjects with COPD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and tolerability of the combination of GSK573719 (500mcg) Inhalation Powder and GW642444 (25mcg) Inhalation Powder administered once-daily via a novel dry powder inhaler (Novel DPI) over 28 days in subjects with COPD

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated written informed consent prior to study participation
* Males or females of non-childbearing potential
* 40 or more years of age
* COPD diagnosis
* 10 pack-years history or greater of cigarette smoking
* Post-bronchodilator FEV1/FVC ratio of 0.70 or less
* Post-bronchodilator FEV1 of 80% or less of predicted normal

Exclusion Criteria:

* Current diagnosis of asthma
* Other significant respiratory disorders besides COPD, including alpha-1 deficiency
* Previous lung resection surgery
* Significant abnormalities in chest x-ray presentation
* Use of oral steroids, antibiotics or hospitalization for a COPD exacerbation within 3 motnhs prior screening
* Any significant disease that would put subject at risk through study participation
* BMI greater than 35
* Pacemaker
* Significantly abnormal ECG, Holter, or clinical lab finding (including Hepatitis B or C)
* Cancer
* Allergy or hypersensitivity to anticholinergics or inhaler excipients
* Diseases that would contra-indicate the use of anticholinergics
* Use of oral corticosteroids within 6 weeks of screening
* Use of long-acting beta-agonists within 48 hours of screening
* Use of tiotropium within 14 days of screening
* Use of theophyllines or anti-leukotrienes within 48 hours of screening
* Use of short-acting bronchodilators within 4 hours of screening
* Use of investigational medicines within 30 days of screening
* Use of high dose inhaled corticosteroids
* Use of long-term oxygen therapy, CPAP or NIPPV
* Previous use of GSK573719 or GW642444

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-01-01; Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Chester, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greenwood, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Feldman G, Walker RR, Brooks J, Mehta R, Crater G. 28-Day safety and tolerability of umeclidinium in combination with vilanterol in COPD: a randomized placebo-controlled trial. Pulm Pharmacol Ther. 2012 Dec;25(6):465-71. doi: 10.1016/j.pupt.2012.08.007. Epub 2012 Aug 31. PMID 22955035
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113120 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113120 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113120 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113120 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113120 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113120 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113120 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria at Screening (Visit 1) completed a 5- to 8-day Run-in period and were then randomized to a 4-week treatment period. A total of 77 par. were screened; 52 par. were randomized and 51 par. received at least one dose of study drug (one par. was randomized in error but did not receive study drug).
Groups:
- Placebo: Participants received matching placebo once daily (QD) via a dry powder inhaler (DPI) in the morning for 4 weeks.
- UMEC/VI 500/25 µg QD: Participants received umeclidinium bromide/vilanterol (UMEC/VI) 500/25 micrograms (µg) QD via a DPI in the morning for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | UMEC/VI 500/25 µg QD
Started | 9 | 42
Completed | 9 | 35
Not Completed | 0 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo QD via a DPI in the morning for 4 weeks.
- UMEC/VI 500/25 µg QD: Participants received UMEC/VI 500/25 µg QD via a DPI in the morning for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC/VI 500/25 µg QD | Total
Number analyzed (Participants) | 9 | 42 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (9.77) | 59.2 (9.48) | 59.1 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 18 | 20
  Male | 7 | 24 | 31
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 6 | 7
  White | 8 | 36 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted Mean Pulse Rate Over 0 to 6 Hours Post-dose at Day 28
Description: Pulse rate is defined as the number of heartbeats in a minute. The weighted mean pulse rate was derived by calculating the area under the pulse rate/time curve (AUC), and then dividing the value by the time interval over which the AUC was calculated. The weighted mean pulse rate was calculated using the 0 to 6 hours post dose measurements at Day 28, which included pre-dose, and post-dose 15 minutes, 45 minutes, 1.5 hours, 3 hours and 6 hours. Baseline pulse rate is the most recent result taken on or before pre-dose Day 1. Change from Baseline is the weighted mean pulse rate at Day 28 minus the Baseline value. Analysis was performed using a repeated measures model with covariates of Baseline pulse rate, sex, age, smoking status, treatment and day and day by treatment and day by Baseline interactions.
Time Frame: Baseline and Day 28
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received >= 1 dose of randomized study medication. All participants with >=1 post-BL assessment and non-missing covariate data are included in the analysis. The number of participants represents participants who provided data at Day 28.
Measure: Least Squares Mean (Standard Error); unit: Beats per minutes (bpm)
Arm/Group | Placebo | UMEC/VI 500/25 µg QD
Number analyzed (Participants) | 9 | 35
Beats per minutes (bpm) | 1.4 (2.20) | 0.9 (1.05)
Statistical Analysis 1: Comparison: Placebo vs UMEC/VI 500/25 µg QD; Test type: Non-Inferiority or Equivalence — UMEC/VI will be declared non-inferior to placebo in terms of weighted mean pulse rate if the upper limit of the 95% confidence interval around the estimated treatment difference for weighted mean pulse rate is less than the non-inferiority margin of +10bpm; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-5.5 to 4.5] — Estimated from repeated measures analysis of covariance

2. Secondary Outcome: Change From Baseline in Weighted Mean Pulse Rate Over 0 to 6 Hours Post-dose at Day 1 and Day 14
Description: Pulse rate is defined as the number of heartbeats in a minute. The weighted mean pulse rate was derived by calculating the area under the pulse rate/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The weighted mean pulse rate was calculated using the 0 to 6 hours post dose measurements on Day 1 and Day 14, which included pre-dose, and post-dose 15 minutes, 45 minutes, 1.5 hours, 3 hours and 6 hours. Baseline pulse rate is the most recent result taken on or before pre-dose Day 1. Change from Baseline is the weighted mean pulse rate at Day 1 or Day 14 minus the Baseline value. Analysis was performed using a repeated measures model with covariates of Baseline pulse rate, sex, age, smoking status, treatment and day and day by treatment and day by Baseline interactions.
Time Frame: Baseline, Day 1, and Day 14
Population: ITT Population. All participants with >=1 post-BL assessment are included in the analysis. Different participants may have been analyzed at different time points (represented by n=X, X in the category titles), so the overall number of participants analyzed reflects everyone in the ITT Population with data avaialable at >=1 time point.
Measure: Least Squares Mean (Standard Error); unit: Beats per minutes
Arm/Group | Placebo | UMEC/VI 500/25 µg QD
Number analyzed (Participants) | 9 | 42
Beats per minutes
  Day 1, n=9, 42 | -1.2 (2.04) | -0.6 (0.92)
  Day 14, n=9, 39 | -1.7 (2.70) | 3.1 (1.26)

3. Secondary Outcome: Change From Baseline in Maximum and Minimum Pulse Rate 0 to 6 Hours Post-dose on Days 1, 14, and 28
Description: Pulse rate is defined as the number of heartbeats in a minute (m). A maximum post-Baseline pulse rate was derived as the maximum value recorded at Days 1, 14 and 28. A minimum post-Baseline pulse rate was derived as the minimum value recorded at Days 1, 14 and 28. The maximum and minimum pulse rates were calculated using the 0 to 6 hours (h) post dose measurements on Days 1, 14 and 28, which included pre-dose, and post-dose 15 m, 45 m, 1.5 h, 3 h and 6 h. Maximum and minimum post-Baseline rate were calculated using the nominal 0-6 h post-dose records, and only records collected during the actual 0-7 h post-dose interval were used. Baseline pulse rate is the most recent result taken on or before pre-dose Day 1. Change from Baseline is the maximum or minimum pulse rate minus the Baseline value. Analysis performed using a repeated measures model with covariates of Baseline pulse rate, sex, age, smoking status, treatment and day and day by treatment and day by Baseline interactions.
Time Frame: Baseline, Day 1, Day 14 and Day 28
Population: ITT Population. The overall number of participants presented is the number who provided at least one post-Baseline assessment of 0-6 hours maximum or minimum pulse rate. Those participants who provided data at the indicated time point are represented by n=X, X in the category titles.
Measure: Least Squares Mean (Standard Error); unit: Beats per minutes
Arm/Group | Placebo | UMEC/VI 500/25 µg QD
Number analyzed (Participants) | 9 | 42
Beats per minutes
  Maximum pulse rate, Day 1, n=9, 42 | 4.5 (2.53) | 6.4 (1.15)
  Maximum pulse rate, Day 14, n=9, 40 | 4.9 (2.93) | 9.7 (1.37)
  Maximum pulse rate, Day 28, n=9, 35 | 7.4 (2.45) | 6.1 (1.19)
  Minimum pulse rate, Day 1, n=9, 42 | -7.0 (2.10) | -6.7 (0.95)
  Minimum pulse rate, Day 14, n=9, 40 | -7.2 (2.78) | -3.2 (1.28)
  Minimum pulse rate, Day 28, n=9, 35 | -6.8 (2.37) | -5.1 (1.15)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication up to 4 weeks.
Description: On-treatment SAEs and non-serious AEs were reported for members of the ITT Population, comprised of all participants who were randomized to treatment and who had received at least one dose of study medication.
Arm/Group | Placebo | UMEC/VI 500/25 µg QD
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/42
Other Adverse Events (participants affected / at risk) | 1/9 | 1/42
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | UMEC/VI 500/25 µg QD (N=42)
Sinusitis (Infections and infestations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.